CLINICAL TRIAL: NCT01373294
Title: Immune Modulation by Addition of Oral Lenalidomide to Intravesical BCG (Bacille Calmette-Guerrin) for Therapy of Non-muscle-invasive Transitional Cell Bladder Cancer
Brief Title: Oral Lenalidomide and Intravesical BCG for Therapy of Bladder Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: H. Lee Moffitt Cancer Center and Research Institute (Other)
Collaborators: Celgene Corporation (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MCC-16295; RV-BLD-PI-0330 (Other: Celgene Corp.)
Record Dates: First submitted 2011-06-13; First posted 2011-06-14 (Estimated); Results first posted 2016-05-12 (Estimated); Last update posted 2019-08-06 (Actual); Status verified 2019-08

CONDITIONS: Bladder Cancer
Keywords: non-muscle-invasive; transitional cell; oral lenalidomide; intravesical
MeSH Terms: conditions — Urinary Bladder Neoplasms | interventions — BCG Vaccine; Lenalidomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- A: Combination Arm (Experimental): Bacille Calmette-Guerrin (BCG) and lenalidomide.
  Participants were assigned to receive BCG or BCG and lenalidomide based on their cancer. This group received BCG + lenalidomide)
  Interventions: Drug: Bacille Calmette-Guerrin (BCG); Drug: Lenalidomide
- B: Control Arm (Active Comparator): Bacille Calmette-Guerrin (BCG) only.
  Participants were assigned to receive BCG or BCG and lenalidomide based on their cancer.
  This group was not eligible to receive the combination of BCG + lenalidomide.
  Interventions: Drug: Bacille Calmette-Guerrin (BCG)

INTERVENTIONS:
Drug: Bacille Calmette-Guerrin (BCG) — Participants will receive BCG instillations once per week for the first 6 weeks. At 3 months and 6 months, participants will receive BCG instillations once per week for three weeks.
  Other Names: BCG Vaccine
Drug: Lenalidomide — Participants may also receive capsules of lenalidomide 10 mg to swallow once per day for 7 months. The study doctor will tell participants if they will be taking lenalidomide.
  Other Names: Revlimid®
  Arms: A: Combination Arm

SUMMARY:
The purposes of this study are to:

* find out whether participants' cancer returns or gets worse while they are taking lenalidomide and Bacille Calmette-Guerrin (BCG);
* evaluate the safety and tolerability of the combination of lenalidomide and BCG;
* compare the cancer progression of participants taking lenalidomide and BCG versus participants taking only BCG

DETAILED DESCRIPTION:
Investigators planned to screen approximately 100 people with bladder cancer who are 18 years of age or older throughout the United States for this study.

This is a multi-center study combining two marketed drugs, one of which has not been used previously in people with transitional cell cancer. Lenalidomide (Revlimid®) is a drug that alters the immune system and it may also interfere with the development of tiny blood vessels that help support tumor growth. Therefore, in theory, it may reduce or prevent the growth of cancer cells. Lenalidomide is approved by the U.S. Food and Drug Administration (FDA) for the treatment of specific types of myelodysplastic syndrome (MDS) and in combination with dexamethasone for patients with multiple myeloma (MM) who have received at least 1 prior therapy. MDS and MM are cancers of the blood. Lenalidomide is currently being tested in a variety of cancer conditions. It is not approved by the FDA for use in people with bladder cancer, so in this case it is considered experimental.

The other drug used in this study is Bacille Calmette-Guerrin (BCG). BCG is approved by the FDA for use in people with bladder cancer.

ELIGIBILITY:
Inclusion Criteria - Either control group or combination treatment:

* Understand and voluntarily sign an informed consent form
* Able to adhere to the study visit schedule and other protocol requirements
* Ta high grade, T1 high grade or Tis transitional cell bladder cancer, s/p transurethral resection of bladder tumor (TURBT) with no remaining resectable disease
* Adequate cardio-pulmonary function (</= Class II ) as defined by New York Heart Association Classification, at the time of screening, and no history of myocardial infarction or heart failure within 6 months of start
* Laboratory test results within these ranges:

  * Absolute neutrophil count ≥ 1500/mm³
  * Platelet count ≥ 75,000
  * Serum creatinine for which computed creatinine clearance is ≥ 30 ml/min, or directly measured creatinine clearance ≥ 30 ml/min
  * Total bilirubin ≤ 1.5 mg/dL
  * Aspartate transaminase (AST) [serum glutamic oxaloacetic transaminase (SGOT)] and Alanine transaminase (ALT) [serum glutamate pyruvic transaminase (SGPT)] ≤ 2 x upper limit of normal (ULN)
* Eastern Cooperative Oncology Group (ECOG) Performance Status of 0, 1 or 2

Inclusion Criteria - Combination treatment:

* Prior BCG treatment for non-muscle invasive transitional cell carcinoma (TCC) last administered < 2 years for Ta high-grade, T1 high grade, Cis, or combination thereof
* Must be registered into the mandatory RevAssist® program, and be willing and able to comply with the requirements of RevAssist®
* Females of childbearing potential (FCBP)† must have a negative serum or urine pregnancy test with a sensitivity of at least 50 mIU/mL within 10 - 14 days prior to and again within 24 hours of starting lenalidomide and must either commit to continued abstinence from heterosexual intercourse or begin TWO acceptable methods of birth control, one highly effective method and one additional effective method AT THE SAME TIME, at least 28 days before she starts taking lenalidomide. FCBP must also agree to ongoing pregnancy testing. Men must agree to use a latex condom during sexual contact with a FCBP even if they have had a successful vasectomy.
* Able to take aspirin (81 or 325 mg) daily as prophylactic anticoagulation (patients intolerant to aspirin may use warfarin or low molecular weight heparin.

Exclusion Criteria:

* Any serious medical condition, laboratory abnormality, or psychiatric illness that would prevent the participant from providing informed consent
* Pregnant or breast feeding (lactating females must agree not to breast feed while taking lenalidomide)
* Any condition, including the presence of laboratory abnormalities, which places the patient at unacceptable risk if he/she were to participate in the study or confounds the ability to interpret data from the study
* Use of any other experimental drug or therapy within 28 days of baseline
* Known hypersensitivity to thalidomide
* Known hypersensitivity to BCG or tuberculosis vaccination
* The development of erythema nodosum if characterized by a desquamating rash while taking thalidomide or similar drugs
* Any prior use of lenalidomide
* Concurrent use of other anti-cancer agents or treatments.
* Known presence of autoimmune disease or immune deficit or chronic disease such as HIV, infectious hepatitis (type B or C), or tuberculosis
* T2+, or N1+, or M+ disease
* Ta or T1 low grade disease only
* Concurrent use of chronic oral steroids, for any indication
* Recent history of deep venous thrombosis currently receiving anticoagulation therapy, with the clot event being in the last 6 months
* Diagnosis of any prior malignancies for the last 5 years with exception of definitively treated basal cell, squamous cell carcinoma of the skin, or carcinoma in-situ of the cervix or breast
* Life expectancy less than 1 year, by treating physician estimate
* Known exposure to person with active tuberculosis within 48 hours of starting treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2011-11-30 (Actual); Primary Completion 2015-01-09 (Actual); Study Completion 2018-12-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mayer Fishman, M.D., Ph.D., Principal Investigator — H. Lee Moffitt Cancer Center and Research Institute
Locations (1):
- H. Lee Moffitt Cancer Center and Research Institute, Tampa, Florida, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Moffitt Cancer Center recruited participants between November 2011 and September 2014.
Pre-assignment Details: Participants were assigned to receive BCG or BCG and lenalidomide based on their cancer.
Groups:
- A: Combination Arm: Bacille Calmette-Guerrin (BCG) and lenalidomide.
- B: Control Arm: Bacille Calmette-Guerrin (BCG).
Period: Overall Study
Arm/Group | A: Combination Arm | B: Control Arm
Started | 15 | 2
Completed | 14 | 2
Not Completed | 1 | 0
Not completed — Adverse Event | 1 | 0

BASELINE CHARACTERISTICS:
Population: The Primary Outcome Measure addresses Arm A only, whose participants received the experimental drug. Too few participants were enrolled into Arm B to conduct the planned per arm comparison. Demographic details and Adverse Events have been reported for all participants in both arms.
Groups:
- Total: Total of all reporting groups
Arm/Group | A: Combination Arm | B: Control Arm | Total
Number analyzed (Participants) | 15 | 2 | 17
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 3 | 0 | 3
  >=65 years | 12 | 2 | 14
Age, Continuous [Mean (Full Range); unit: years] | 72 [52 to 85] | 70 [66 to 74] | 71.8 [52 to 85]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 0 | 1
  Male | 14 | 2 | 16
Region of Enrollment [Number; unit: participants]
  United States | 15 | 2 | 17

OUTCOME MEASURES:

1. Primary Outcome: Arm A: Progression Free Survival (PFS)
Description: The 1-year progression free/ recurrence free/ bladder-intact survival was tabulated for the experimental arm for a median follow-up period of 369 days. The progression free/ recurrence free/ bladder-intact survival is defined as the time from start of study treatment to first documentation of objective tumor progression, recurrence, bladder resection or irradiation or to death due to any cause, whichever comes first. PFS data was not collected for participants in the Arm B: Control because too few participants were enrolled in Arm B to conduct the planned per Arm comparison
Time Frame: 1 year
Population: Experimental Arm A Group Only.
Measure: Number; unit: participants
Arm/Group | A: Combination Arm
Number analyzed (Participants) | 15
participants | 8

2. Secondary Outcome: Treatment Emergent Adverse Events (AEs) or Serious Adverse Events (SAEs)
Description: Number of participants with treatment emergent AEs or SAEs per category. SAEs will be specifically labeled as such. Participants were assessed at monthly intervals (corresponding to Revlimid™ refill points for adverse events), classified by Common Terminology Criteria for Adverse Events (CTCAE) version 4.0, and these were tabulated.
Time Frame: Duration of study treatment and follow-up - average of 12 months
Population: All participants.
Measure: Number; unit: participants
Arm/Group | A: Combination Arm | B: Control Arm
Number analyzed (Participants) | 15 | 2
participants
  Hematuria | 6 | 1
  Urinary frequency | 3 | 0
  Urinary urgency | 3 | 1
  Urinary tract pain | 2 | 0
  Bladder spasm | 1 | 0
  Fatigue | 7 | 0
  Edema face | 1 | 0
  Edema limbs | 1 | 0
  Fever | 1 | 0
  Pain | 1 | 0
  Nausea | 2 | 0
  Erythroderma | 1 | 0
  Pruritus | 1 | 0
  Rash acneiform | 1 | 0
  Rash maculo-papular | 1 | 0
  Urinary tract infection | 2 | 0
  Pharyngitis | 1 | 0
  Platelet count decreased | 1 | 0
  SAE: Grade 3 Myocardial infarction | 1 | 0
  Headache | 1 | 0
  Peripheral sensory neuropathy | 1 | 0

3. Other Pre Specified Outcome: Effect of Addition of Revlimid on Cytokines
Description: The immunologic impact of the addition of Revlimid™ to BCG for secondary prevention of non-muscle-invasive transitional cell bladder cancer, in terms of a panel of correlative assays. The effect of addition of Revlimid on cytokines associated with generation of immune response and on cytotoxic T lymphocytes and memory phenotype lymphocytes.
Time Frame: Duration of study treatment and follow-up - average of 12 months
Reporting Status: Not Posted

4. Other Pre Specified Outcome: Comparison of the Correlative Assay
Description: For comparing the correlative assay results of ever-relapsers vs non-relapsers, the combined data with the monotherapy and combination therapy groups would be applied. The participants would be categorized based on 1-year relapse.
Time Frame: 1 year post disease response
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 36 months
Arm/Group | A: Combination Arm | B: Control Arm
Serious Adverse Events (participants affected / at risk) | 2/15 | 0/2
Other Adverse Events (participants affected / at risk) | 15/15 | 1/2
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | A: Combination Arm (N=15) | B: Control Arm (N=2)
Myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | A: Combination Arm (N=15) | B: Control Arm (N=2)
Hematuria (Renal and urinary disorders) | 7 (9) | 0 (0)
Urinary frequency (Renal and urinary disorders) | 3 (5) | 0 (0)
Urinary urgency (Renal and urinary disorders) | 3 (3) | 0 (0)
Urinary tract pain (Renal and urinary disorders) | 2 (3) | 0 (0)
Bladder spasm (Renal and urinary disorders) | 1 (1) | 0 (0)
Urinary incontinence (Renal and urinary disorders) | 0 (0) | 1 (1)
Fatigue (General disorders) | 7 (9) | 0 (0)
Edema face (General disorders) | 1 (1) | 0 (0)
Edema limbs (General disorders) | 1 (1) | 0 (0)
Fever (General disorders) | 1 (2) | 0 (0)
Pain (General disorders) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 3 (5) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 3 (3) | 0 (0)
Nausea (Gastrointestinal disorders) | 2 (2) | 0 (0)
Gastrointestinal disorders - Other, soreness over suprapubic area (Gastrointestinal disorders) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 3 (4) | 0 (0)
Pharyngitis (Infections and infestations) | 1 (1) | 0 (0)
Erythroderma (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Rash acneiform (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Weight loss (Investigations) | 2 (2) | 0 (0)
Platelet count decreased (Investigations) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Atrial flutter (Cardiac disorders) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 0 (0)
Peripheral sensory neuropathy (Nervous system disorders) | 1 (2) | 0 (0)
Anxiety (Psychiatric disorders) | 1 (1) | 0 (0)
Depression (Psychiatric disorders) | 1 (1) | 0 (0)
Blood and lymphatic system disorders - Other, blood clots in urine (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
This study closed to accrual early, due to slow accrual. Too few participants were enrolled into Arm B to conduct the planned per arm comparisons.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes